CLINICAL TRIAL: NCT04155736
Title: A Randomized Controlled Trial of a Self-Management App for Symptoms of Posttraumatic Stress: The Role of Coaching Support
Brief Title: Testing a Self-Management App for Symptoms of Posttraumatic Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52829
Record Dates: First submitted 2019-10-30; First posted 2019-11-07 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Renew with coaching (Experimental): Users will be assigned a study staff member as a support person who is notified when the user engages with the app or if they have not engaged for 7 days. Support persons are provided with psychoeducation material including information about how to be an effective support person for the user and direct messaging capacity to respond to app notifications about user engagement (e.g., user earned X points, user achieved a new level).
  Interventions: Behavioral: Renew
- Renew without coaching (Active Comparator): Same as "Renew with coaching" except that the users will not be assigned a study staff member as a support person.
  Interventions: Behavioral: Renew
- Wait list (No Intervention): No intervention is provided

INTERVENTIONS:
Behavioral: Renew — Renew is a behavioral health self-management app/too that focuses on three core activities: 1) in vivo exposure (to help participants approach safe situations they have been avoiding that they want to feel comfortable in), 2) expressive writing (to help participants emotionally process trauma memories), and 3) Self-Care exercises (designed to promote behavioral activation, social connectedness and relaxation; includes a breathing relaxation tool). Users have access to psychoeducation via a whiteboard video and short texts as well as Motivation content (quotes, videos, images, and songs) related to confronting challenges and overcoming fears. For each exercise that is completed, the user earns points that are connected to levels and visually reinforcing images (i.e., a growing tree).
  Arms: Renew with coaching; Renew without coaching

SUMMARY:
The purpose of this study is to evaluate the acceptability and efficacy of a self-guided behavioral health tool delivered by mobile app (called "Renew") for people who are experiencing symptoms of posttraumatic stress. This study also aims to determine the necessity of coaching support over and above support from peers, shedding light on the critical question of level of support resources needed to maintain mHealth app engagement.

ELIGIBILITY:
Inclusion Criteria:

* Veterans 18 years or older
* own an Android smart phone (as the app is only available for Android)
* self-report having experiencing symptoms of posttraumatic stress (defined as a PCL-5 score of 31 or higher).

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-07-11 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2021-02-06 (Actual)

PRIMARY OUTCOMES:
Post Traumatic Stress Disorder CheckList for Diagnostic and Statistical Manual - 5 (PCL-5; Weathers, et al., 2013) | Approximately 10-weeks after participant enrollment
  Self report measure of PTSD symptoms. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. Higher scores indicate greater PTSD severity.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer, & Williams, 2001) | Approximately 10-weeks after participant enrollment
  Self report measure of depression symptoms. It is the 9-item measure that yields a total score of 0-27, with higher scores indicating greater depressive symptom severity.
A PTSD coping self-efficacy measure, developed following Bandura's (2006) guidelines | Approximately 10-weeks after participant enrollment
  Self report measure of PTSD coping self-efficacy. It is a 10-item measure that yields a total score of 0-1000, with higher scores indicating greater coping self-efficacy.
Multidimensional Scale of Perceived Social Support (Zimet, Dahlem, Zimet, & Farley, (1988) | Approximately 10-weeks after participant enrollment
  Self report measure of perceived social support. It is a 12-item measure that yields a total score of 12-84, with higher scores indicating greater perceived social support.
Perceived helpfulness of Renew | Approximately 6-weeks after participant enrollment
  Phone interview to assess perceived helpfulness of Renew. This is a qualitative measure.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen McLean, PhD, Principal Investigator — Palo Alto Veterans Institute for Research
Locations (1):
- VA Palo Alto Healthcare System, Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McLean C, Davis CA, Miller M, Ruzek J, Neri E. The Effects of an Exposure-Based Mobile App on Symptoms of Posttraumatic Stress Disorder in Veterans: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2022 Nov 4;10(11):e38951. doi: 10.2196/38951. PMID 36331540